CLINICAL TRIAL: NCT00853749
Title: REVACCINATION WITH PREVENAR 13 - CHARACTERIZATION OF THE LATE IMMUNE RESPONSE AFTER POLYSACCHARIDE (REPLAY).
Brief Title: Immune Response In Children Revaccinated With Pneumococcal Conjugate Vaccine
Acronym: REPLAY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Masking: None | Purpose: Other
Other Study IDs: 6096A1-3013; B1851012 (Other: Alias Study Number); 2008-006194-33 (EudraCT Number)
Record Dates: First submitted 2009-02-19; First posted 2009-03-02 (Estimated); Results first posted 2011-01-05 (Estimated); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Invasive Pneumococcal Disease
Keywords: Immune response; pneumococcal conjugate vaccine; polysaccharide
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single (Other): All subjects will receive a single dose of 13vPnC
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine (13vPnC); Procedure: Blood draw

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine (13vPnC) — 0.5 mL intramuscular injection
Procedure: Blood draw — Collection of 10 mL of blood

SUMMARY:
The primary purpose of this study is to evaluate the immune response to 13-valent pneumococcal conjugate vaccine (13vPnCV) in children who as infants received either a complete series of PnCV versus a combination of PnCV and pneumococcal polysaccharide vaccine (PSV). This study is also intended to evaluate the safety of the 13vPnC.

DETAILED DESCRIPTION:
Follow-up measure for the EMEA supporting a Type II variation for Prevenar (PCV7) label

ELIGIBILITY:
Inclusion Criteria:

* Fully vaccinated children who participated in a previous Wyeth study (Study D139-P506) and received a booster dose of either 23-valent pneumococcal polysaccharide vaccine (PPV23) or pneumococcal conjugate vaccine (PnCV) per the original protocol for that study.
* Subjects must be in good health as determined by medical history, physical examination and clinical judgment.

Exclusion Criteria:

* Known allergy to any component of the 7-valent pneumococcal conjugate vaccine (7vPnC) or 13-valent pneumococcal conjugate vaccine (13vPnC).
* History of documented invasive pneumococcal disease (defined as a positive culture of S. pneumoniae from a normally sterile body site).
* Any known or suspected disease or dysfunction of the immune system, including: HIV infection, Malignancy, Receipt of immunosuppressive therapy, Sickle cell hemoglobinopathy.
* Receipt of immune-globulin within the past 3 months.
* Receipt of either PSV or 7vPnCV since the completion of Study D139-P506.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 89 (Actual)
Dates: Start 2009-05-05 (Actual); Primary Completion 2009-12-16 (Actual); Study Completion 2009-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Iceland (2):
  - Landspitali University Hospital, Hringbraut, Reykjavik
  - Midstod Heilsuverndar barna, Reykjavik

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Sigurdardottir ST, Center KJ, Davidsdottir K, Arason VA, Hjalmarsson B, Elisdottir R, Ingolfsdottir G, Northington R, Scott DA, Jonsdottir I. Decreased immune response to pneumococcal conjugate vaccine after 23-valent pneumococcal polysaccharide vaccine in children. Vaccine. 2014 Jan 9;32(3):417-24. doi: 10.1016/j.vaccine.2013.11.029. Epub 2013 Dec 2. PMID 24300594
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6096A1-3013&StudyName=Immune%20Response%20In%20Children%20Revaccinated%20With%20Pneumococcal%20Conjugate%20Vaccine

RESULTS

PARTICIPANT FLOW:
Groups:
- PCV/23vPS/13vPnC: For this study, participants received a single 0.5 milliliter (mL) dose of 13-valent pneumococcal conjugate vaccine (13vPnC), administered intramuscularly. Participants previously must have also received an infant series of 9-valent pneumococcal-conjugate-meningococcal serogroup C conjugate combination vaccine (9V-MnCC) also known as pneumococcal conjugate vaccine (PCV) followed by a toddler dose of 23-valent pneumococcal polysaccharide vaccine (23vPS).
- PCV/PCV/13vPnC: For this study, participants received a single 0.5 mL dose of 13vPnC administered intramuscularly. Participants must have also previously received 9V-MnCC followed by a toddler dose of 9V-MnCC (also referred to as PCV).
Period: Overall Study
Arm/Group | PCV/23vPS/13vPnC | PCV/PCV/13vPnC
Started | 50 | 39
Vaccinated | 50 | 39
Completed | 50 | 38
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCV/23vPS/13vPnC | PCV/PCV/13vPnC | Total
Number analyzed (Participants) | 50 | 39 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (0.2) | 7.6 (0.2) | 7.6 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 45
  Male | 25 | 19 | 44

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Predefined Serotype-specific Immunoglobulin G (IgG) Antibody Concentration Greater Than or Equal to ( ≥) 0.35 Micrograms Per Milliliter (mcg/mL) Measured 1 Month After Vaccination
Description: Percentage of participants achieving predefined antibody threshold ≥ 0.35 mcg/mL along with the corresponding 95 percent (%) Confidence Interval (CI) for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: Day 28
Population: Evaluable Immunogenicity Population: received 1 dose of 13vPnC at Visit 1, blood drawn within specified timeframes, at least 1 valid and determinate assay result at Visits 1 and 3, no major protocol violations, and no prohibited vaccines. N=number of participants with a determinate IgG antibody concentration to the given serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PCV/23vPS/13vPnC | PCV/PCV/13vPnC
Number analyzed (Participants) | 50 | 37
Percentage of participants
  Common Serotype 4 | 100.0 [92.9 to 100.0] | 97.3 [85.8 to 99.9]
  Common Serotype 6B | 100.0 [92.9 to 100.0] | 100.0 [90.5 to 100.0]
  Common Serotype 9V | 100.0 [92.9 to 100.0] | 100.0 [90.5 to 100.0]
  Common Serotype 14 | 100.0 [92.7 to 100.0] | 100.0 [90.5 to 100.0]
  Common Serotype18C | 100.0 [92.9 to 100.0] | 97.3 [85.8 to 99.9]
  Common Serotype 19F | 100.0 [92.9 to 100.0] | 100.0 [90.5 to 100.0]
  Common Serotype 23F | 100.0 [92.9 to 100.0] | 100.0 [90.5 to 100.0]
  Additional Serotype 1 | 100.0 [92.9 to 100.0] | 97.3 [85.8 to 99.9]
  Additional Serotype 3 | 100.0 [92.9 to 100.0] | 100.0 [90.5 to 100.0]
  Additional Serotype 5 | 100.0 [92.9 to 100.0] | 100.0 [90.5 to 100.0]
  Additional Serotype 6A | 100.0 [92.9 to 100.0] | 100.0 [90.5 to 100.0]
  Additional Serotype 7F | 100.0 [92.9 to 100.0] | 100.0 [90.5 to 100.0]
  Additional Serotype 19A | 100.0 [92.9 to 100.0] | 100.0 [90.5 to 100.0]
Statistical Analysis 1: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 4; Test type: Superiority or Other; Difference in proportions (percentage) = 2.7, 95% CI 2-sided [-5.0 to 14.2]
Statistical Analysis 2: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 6B; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.3 to 9.5]
Statistical Analysis 3: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 9V; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.3 to 9.5]
Statistical Analysis 4: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 14; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.8 to 9.5]
Statistical Analysis 5: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 18C; Test type: Superiority or Other; Difference in proportions (percentage) = 2.7, 95% CI 2-sided [-5.0 to 14.2]
Statistical Analysis 6: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 19F; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.3 to 9.5]
Statistical Analysis 7: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 23F; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.3 to 9.5]
Statistical Analysis 8: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for additional serotype 1; Test type: Superiority or Other; Difference in proportions (percentage) = 2.7, 95% CI 2-sided [-5.0 to 14.2]
Statistical Analysis 9: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for additional serotype 3; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.3 to 9.5]
Statistical Analysis 10: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for additional serotype 5; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.3 to 9.5]
Statistical Analysis 11: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for additional serotype 6A; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.3 to 9.5]
Statistical Analysis 12: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for additional serotype 7F; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.3 to 9.5]
Statistical Analysis 13: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for additional serotype 19A; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.3 to 9.5]

2. Primary Outcome: Percentage of Participants Achieving Opsonophagocytic Assay (OPA) Titers ≥ 1:8 Measured 1 Month After Vaccination
Description: Percentage of participants achieving OPA along with the corresponding 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. Exact 2-sided CI based on the observed proportion of participants.
Time Frame: Day 28
Population: Evaluable Immunogenicity Population; N=number of participants with a determinate OPA antibody titer to the given serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | PCV/23vPS/13vPnC | PCV/PCV/13vPnC
Number analyzed (Participants) | 50 | 37
Percentage of participants
  Common Serotype 4 | 98.0 [89.4 to 99.9] | 97.2 [85.5 to 99.9]
  Common Serotype 6B | 100.0 [92.7 to 100.0] | 100.0 [90.3 to 100.0]
  Common Serotype 9V | 100.0 [92.7 to 100.0] | 100.0 [90.3 to 100.0]
  Common Serotype 14 | 100.0 [92.7 to 100.0] | 100.0 [90.3 to 100.0]
  Common Serotype 18C | 100.0 [92.9 to 100.0] | 100.0 [90.0 to 100.0]
  Common Serotype 19F | 100.0 [92.7 to 100.0] | 100.0 [90.0 to 100.0]
  Common Serotype 23F | 98.0 [89.4 to 99.9] | 100.0 [89.7 to 100.0]
  Additional Serotype 1 | 100.0 [92.9 to 100.0] | 97.3 [85.8 to 99.9]
  Additional Serotype 3 | 98.0 [89.1 to 99.9] | 100.0 [90.3 to 100.0]
  Additional Serotype 5 | 98.0 [89.4 to 99.9] | 97.3 [85.8 to 99.9]
  Additional Serotype 6A | 100.0 [92.9 to 100.0] | 100.0 [90.5 to 100.0]
  Additional Serotype 7F | 98.0 [89.4 to 99.9] | 100.0 [90.3 to 100.0]
  Additional Serotype 19A | 100.0 [92.9 to 100.0] | 100.0 [90.5 to 100.0]
Statistical Analysis 1: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 4; Test type: Superiority or Other; Difference in proportions (percentage) = 0.8, 95% CI 2-sided [-8.6 to 12.7]
Statistical Analysis 2: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 6B; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.5 to 9.7]
Statistical Analysis 3: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 9V; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.5 to 9.7]
Statistical Analysis 4: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 14; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.5 to 9.7]
Statistical Analysis 5: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 18C; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.4 to 10.0]
Statistical Analysis 6: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 19F; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.5 to 10.0]
Statistical Analysis 7: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for common serotype 23F; Test type: Superiority or Other; Difference in proportions (percentage) = -2.0, 95% CI 2-sided [-10.8 to 8.1]
Statistical Analysis 8: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for additional serotype 1; Test type: Superiority or Other; Difference in proportions (percentage) = 2.7, 95% CI 2-sided [-5.0 to 14.2]
Statistical Analysis 9: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for additional serotype 3; Test type: Superiority or Other; Difference in proportions (percentage) = -2.0, 95% CI 2-sided [-11.1 to 7.9]
Statistical Analysis 10: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for additional serotype 5; Test type: Superiority or Other; Difference in proportions (percentage) = 0.7, 95% CI 2-sided [-8.5 to 12.2]
Statistical Analysis 11: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for additional serotype 6A; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.3 to 9.5]
Statistical Analysis 12: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for additional serotype 7F; Test type: Superiority or Other; Difference in proportions (percentage) = -2.0, 95% CI 2-sided [-11.3 to 7.7]
Statistical Analysis 13: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for additional serotype 19A; Test type: Superiority or Other; Difference in proportions (percentage) = 0.0, 95% CI 2-sided [-7.3 to 9.5]

3. Secondary Outcome: Antibody Response Measured 1 Month After Vaccination (Avidity Assay)
Description: Avidity assay had measurable range of 0.117 to 7.5. Results expressed as avidity index (AI). Geometric mean avidity presented for 3 common pneumococcal serotypes (serotype 6B, 19F, and 23F) and 2 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1 and 5).
Time Frame: Day 28
Population: Evaluable Immunogenicity Population; In accordance with the recommendation of the lab completing the assays, values above the upper limit were assigned a value of 8.0 and those below the lower limit were assigned a value of 0.10. N=number of participants with a determinate avidity index for the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: AI
Arm/Group | PCV/23vPS/13vPnC | PCV/PCV/13vPnC
Number analyzed (Participants) | 50 | 36
AI
  Additional serotype 1 | 1.42 [1.15 to 1.76] | 4.68 [3.62 to 6.04]
  Additional serotype 5 | 1.85 [1.46 to 2.36] | 5.85 [4.81 to 7.11]
  Common serotype 6B | 2.43 [1.77 to 3.35] | 5.48 [4.38 to 6.86]
  Common serotype 19F | 2.17 [1.69 to 2.79] | 2.46 [1.88 to 3.21]
  Common serotype 23F | 3.02 [2.36 to 3.85] | 6.43 [5.33 to 7.76]
Statistical Analysis 1: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 1: Ratio of geometric mean avidity (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of geometric means = 0.30, 95% CI 2-sided [0.22 to 0.42] — CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures (PCV/23vPS/13vPnC, PCV/PCV/13vPnC)
Statistical Analysis 2: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 5: Ratio of geometric mean avidity (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of geometric means = 0.32, 95% CI 2-sided [0.23 to 0.44] — CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures ((PCV/23vPS/13vPnC, PCV/PCV/13vPnC)
Statistical Analysis 3: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 6B: Ratio of geometric mean avidity (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of geometric means = 0.44, 95% CI 2-sided [0.29 to 0.67] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 19F: Ratio of geometric mean avidity (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of geometric means = 0.88, 95% CI 2-sided [0.61 to 1.27] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 23F: Ratio of geometric mean avidity (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of geometric means = 0.47, 95% CI 2-sided [0.34 to 0.65] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Antibody Response Measured 1 Month After Vaccination (OPA)
Description: Antibody response as measured by OPA, 1 month after vaccination. Geometric mean titers (GMTs) calculated using all participants with available data for the specified blood draw. CIs were back transformations of a CI based on the Student t distribution for the mean logarithm of the titers.
Time Frame: Day 28
Population: Evaluable Immunogenicity Population; N=number of participants with a determinate antibody titre to the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: GMT
Arm/Group | PCV/23vPS/13vPnC | PCV/PCV/13vPnC
Number analyzed (Participants) | 50 | 37
GMT
  Common Serotype 4 | 2374 [1656.3 to 3404.0] | 3765 [2339.1 to 6059.8]
  Common Serotype 6B | 11156 [9073.5 to 13715.2] | 11477 [8418.5 to 15646.8]
  Common Serotype 9V | 1651 [1067.8 to 2553.3] | 1713 [1087.0 to 2700.0]
  Common Serotype 14 | 3041 [2311.4 to 4001.1] | 3048 [2318.3 to 4006.9]
  Common Serotype 18C | 3230 [2616.1 to 3987.1] | 5684 [3122.2 to 10349.6]
  Common Serotype 19F | 1266 [1013.9 to 1582.0] | 1198 [842.3 to 1703.9]
  Common Serotype 23F | 1678 [1212.3 to 2322.1] | 2714 [1970.1 to 3739.5]
  Additional Serotype 1 | 217 [162.6 to 290.5] | 1087 [717.5 to 1646.3]
  Additional Serotype 3 | 153 [117.2 to 200.2] | 188 [146.6 to 240.8]
  Additional Serotype 5 | 264 [178.5 to 389.9] | 719 [500.9 to 1032.4]
  Additional Serotype 6A | 7060 [5352.2 to 9312.6] | 5034 [3336.6 to 7594.4]
  Additional Serotype 7F | 5835 [4160.0 to 8184.1] | 7887 [6447.9 to 9647.0]
  Additional Serotype 19A | 1256 [990.9 to 1591.9] | 1556 [1108.8 to 2182.2]
Statistical Analysis 1: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 4: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 0.6, 95% CI 2-sided [0.35 to 1.12] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 6B: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 1.0, 95% CI 2-sided [0.68 to 1.38] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 9V: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 1.0, 95% CI 2-sided [0.51 to 1.81] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 14: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 1.0, 95% CI 2-sided [0.67 to 1.48] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 18C: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 0.6, 95% CI 2-sided [0.33 to 0.98] — CIs for the ratio were back transformations of a CI based on the Student t distribution for the mean difference of the logarithms of the measures(PCV/23vPS/13vPnC, PCV/PCV/13vPnC)
Statistical Analysis 6: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 19F: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 1.1, 95% CI 2-sided [0.72 to 1.56] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 23F: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 0.6, 95% CI 2-sided [0.39 to 0.99] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 1: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 0.2, 95% CI 2-sided [0.12 to 0.32] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 3: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 0.8, 95% CI 2-sided [0.56 to 1.18] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 5: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 0.4, 95% CI 2-sided [0.21 to 0.63] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 6A: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 1.4, 95% CI 2-sided [0.88 to 2.25] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 7F: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 0.7, 95% CI 2-sided [0.48 to 1.14] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 19A: Ratio of GMTs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMTs = 0.8, 95% CI 2-sided [0.54 to 1.20] — [estimate comment as in outcome 3, analysis 1]

5. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal IgG Antibody 1 Month After Vaccination
Description: Antibody GMC as measured by mcg/mL for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were evaluated. CIs were back transformations of a CI based on the Student t distribution for the mean logarithm of the concentrations. GMCs were calculated using all participants with available data for the specified blood draw.
Time Frame: Day 28
Population: Evaluable Immunogenicity Population; N=number of participants with a determinate antibody concentration to the specified serotype.
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | PCV/23vPS/13vPnC | PCV/PCV/13vPnC
Number analyzed (Participants) | 50 | 37
mcg/mL
  Common serotype 4 | 4.18 [3.38 to 5.16] | 11.34 [7.74 to 16.62]
  Common serotype 6B | 29.51 [21.32 to 40.83] | 41.70 [29.01 to 59.96]
  Common serotype 9V | 4.31 [3.68 to 5.04] | 7.39 [6.05 to 9.03]
  Common serotype 14 | 17.47 [12.76 to 23.93] | 22.78 [15.75 to 32.96]
  Common serotype 18C | 2.76 [2.15 to 3.56] | 4.83 [3.48 to 6.71]
  Common serotype 19F | 9.78 [7.45 to 12.83] | 11.60 [8.46 to 15.92]
  Common serotype 23F | 7.89 [6.18 to 10.07] | 12.25 [8.92 to 16.81]
  Additional serotype 1 | 5.28 [4.22 to 6.61] | 19.43 [13.77 to 27.41]
  Additional serotype 3 | 3.28 [2.44 to 4.41] | 2.87 [2.19 to 3.76]
  Additional serotype 5 | 5.75 [4.64 to 7.12] | 15.98 [11.99 to 21.30]
  Additional serotype 6A | 11.16 [8.80 to 14.16] | 14.07 [10.64 to 18.61]
  Additional serotype 7F | 7.13 [5.67 to 8.96] | 8.05 [5.94 to 10.91]
  Additional serotype 19A | 14.62 [11.49 to 18.59] | 17.07 [12.92 to 22.55]
Statistical Analysis 1: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 4: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 0.37, 95% CI 2-sided [0.25 to 0.55] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 2: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 6B: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 0.71, 95% CI 2-sided [0.44 to 1.15] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 9V: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 0.58, 95% CI 2-sided [0.45 to 0.75] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 14: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 0.77, 95% CI 2-sided [0.48 to 1.24] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 5: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 18C: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 0.57, 95% CI 2-sided [0.38 to 0.85] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 6: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 19F: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 0.84, 95% CI 2-sided [0.56 to 1.27] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 7: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 23F: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 0.64, 95% CI 2-sided [0.44 to 0.95] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 8: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 1: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 0.27, 95% CI 2-sided [0.18 to 0.40] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 9: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 3: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 1.14, 95% CI 2-sided [0.76 to 1.72] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 10: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 5: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 0.36, 95% CI 2-sided [0.25 to 0.51] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 11: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 6A: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 0.79, 95% CI 2-sided [0.55 to 1.14] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 12: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 7F: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 0.89, 95% CI 2-sided [0.61 to 1.28] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 13: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Serotype 19A: Ratio of GMCs (PCV/23vPS/13vPnC, PCV/PCV/13vPnC); Test type: Superiority or Other; Ratio of GMCs = 0.86, 95% CI 2-sided [0.60 to 1.23] — [estimate comment as in outcome 3, analysis 1]

6. Other Pre Specified Outcome: Percentage of Participants Reporting Prespecified Local Reactions Within 4 Days of Vaccination
Description: Local reactions were reported by the parent/legal guardian using a diary card. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Redness and swelling were scaled as Any (redness or swelling present); Mild (0.5 centimeters [cm] to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may have been represented in more than 1 category.
Time Frame: Day 1 through Day 4
Population: Safety Population: all participants who receive at least 1 dose of the study vaccine; N=number of participants reporting yes for at least 1 day or no for all days and "number analyzed" signifies participants reporting the specific characteristic.
Measure: Number; unit: Percentage of participants
Arm/Group | PCV/23vPS/13vPnC | PCV/PCV/13vPnC
Number analyzed (Participants) | 50 | 39
Percentage of participants
  Tenderness: Any: number analyzed (Participants) | 44 | 30
  Tenderness: Any | 88.0 | 76.9
  Tenderness: Significant: number analyzed (Participants) | 6 | 8
  Tenderness: Significant | 12.0 | 20.5
  Redness: Any: number analyzed (Participants) | 25 | 26
  Redness: Any | 50.0 | 66.7
  Redness: Mild: number analyzed (Participants) | 5 | 6
  Redness: Mild | 10.0 | 15.8
  Redness: Moderate: number analyzed (Participants) | 20 | 20
  Redness: Moderate | 40.0 | 52.6
  Redness: Severe: number analyzed (Participants) | 5 | 8
  Redness: Severe | 10.0 | 21.1
  Swelling: Any: number analyzed (Participants) | 22 | 23
  Swelling: Any | 44.0 | 59.0
  Swelling: Mild: number analyzed (Participants) | 8 | 10
  Swelling: Mild | 16.3 | 26.3
  Swelling: Moderate: number analyzed (Participants) | 14 | 17
  Swelling: Moderate | 28.6 | 44.7
  Swelling: Severe: number analyzed (Participants) | 1 | 3
  Swelling: Severe | 2.0 | 7.9
Statistical Analysis 1: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for any tenderness; Test type: Superiority or Other; p = 0.253, Fisher Exact
Statistical Analysis 2: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for significant tenderness; Test type: Superiority or Other; p = 0.380, Fisher Exact
Statistical Analysis 3: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for any redness; Test type: Superiority or Other; p = 0.135, Fisher Exact
Statistical Analysis 4: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for mild redness; Test type: Superiority or Other; p = 0.520, Fisher Exact
Statistical Analysis 5: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for moderate redness; Test type: Superiority or Other; p = 0.283, Fisher Exact
Statistical Analysis 6: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for severe redness; Test type: Superiority or Other; p = 0.225, Fisher Exact
Statistical Analysis 7: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for any swelling; Test type: Superiority or Other; p = 0.202, Fisher Exact
Statistical Analysis 8: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for mild swelling; Test type: Superiority or Other; p = 0.294, Fisher Exact
Statistical Analysis 9: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for moderate swelling; Test type: Superiority or Other; p = 0.175, Fisher Exact
Statistical Analysis 10: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for severe swelling; Test type: Superiority or Other; p = 0.314, Fisher Exact

7. Other Pre Specified Outcome: Percentage of Participants Reporting Prespecified Systemic Reactions Within 4 Days of Vaccination
Description: Pre-specified systemic events (any fever 38 degrees Celsius [C], decreased appetite, irritability, increased sleep, and decreased sleep) were reported using a diary card. Participants may have been represented in more than 1 category.
Time Frame: Day 1 through Day 4
Population: Safety; N=number of participants reporting yes for at least 1 day or no for all days and number analyzed signifies participants reporting the specific characteristic.
Measure: Number; unit: Percentage of participants
Arm/Group | PCV/23vPS/13vPnC | PCV/PCV/13vPnC
Number analyzed (Participants) | 50 | 39
Percentage of participants
  Fever ≥ 38 degrees C but ≤ 39 degrees C: number analyzed (Participants) | 1 | 1
  Fever ≥ 38 degrees C but ≤ 39 degrees C | 2.0 | 2.8
  Decreased appetite: number analyzed (Participants) | 6 | 4
  Decreased appetite | 12.2 | 10.3
  Irritability: number analyzed (Participants) | 9 | 4
  Irritability | 18.4 | 11.4
  Increased sleep: number analyzed (Participants) | 2 | 5
  Increased sleep | 4.0 | 12.8
  Decreased sleep: number analyzed (Participants) | 0 | 2
  Decreased sleep |  | 5.1
  Rash: number analyzed (Participants) | 3 | 1
  Rash | 6.0 | 2.6
Statistical Analysis 1: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for fever ≥ 38 degrees C but ≤ 39 degrees C; Test type: Superiority or Other; p > .99, Fisher Exact
Statistical Analysis 2: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for decreased appetite; Test type: Superiority or Other; p > .99, Fisher Exact
Statistical Analysis 3: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for irritability; Test type: Superiority or Other; p = 0.543, Fisher Exact
Statistical Analysis 4: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for increased sleep; Test type: Superiority or Other; p = 0.233, Fisher Exact
Statistical Analysis 5: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for decreased sleep; Test type: Superiority or Other; p = 0.198, Fisher Exact
Statistical Analysis 6: Comparison: PCV/23vPS/13vPnC vs PCV/PCV/13vPnC; Comparison between treatments for rash; Test type: Superiority or Other; p = 0.628, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline through 1 Month after last study vaccination (28 Days). Local reactions and systemic events assessed within 4 days of dose (Day 1 through Day 4)
Description: The same event may appear as both an adverse event (AE) and a Serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- PCV/23vPS/13vPnC: For this study, participants received a single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC) administered intramuscularly. Participants previously must have also received an infant series of 9-valent pneumococcal-conjugate-meningococcal serogroup C conjugate combination vaccine (9V-MnCC) also known as pneumococcal conjugate vaccine (PCV) followed by a toddler dose of 23-valent pneumococcal polysaccharide vaccine (23vPS).
  Other AEs (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=8; systematic (solicited) Local Reactions N=44; systematic (solicited) Systemic Events N=9.
- PCV/PCV/13vPnC: For this study, participants received a single 0.5 mL dose of 13vPnC, administered intramuscularly. Participants must have also previously received 9V-MnCC followed by a toddler dose of 9V-MnCC (also referred to as PCV).
  Other AEs (non-serious events): the number affected (N) for nonsystematic (unsolicited) Other Adverse Events N=7; systematic (solicited) Local Reactions N=30; systematic (solicited) Systemic Events N=5.
Arm/Group | PCV/23vPS/13vPnC | PCV/PCV/13vPnC
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/39
Other Adverse Events (participants affected / at risk) | 44/50 | 30/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | PCV/23vPS/13vPnC (N=50) | PCV/PCV/13vPnC (N=39)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Viral infection (Infections and infestations) | 0 | 3
Influenza (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Tenderness (Any) (Skin and subcutaneous tissue disorders) | 44 | 30
Tenderness (Significant) (Skin and subcutaneous tissue disorders) | 6 | 8
Redness (Any) (Skin and subcutaneous tissue disorders) | 25 | 26
Redness (Mild) (Skin and subcutaneous tissue disorders) | 5 | 6/38
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 20 | 20/38
Redness (Severe) (Skin and subcutaneous tissue disorders) | 5 | 8/38
Swelling (Any) (Skin and subcutaneous tissue disorders) | 22 | 23
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 8/49 | 10/38
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 14/49 | 17/38
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 1/49 | 3/38
Fever ≥ 38°C but ≤ 39°C (General disorders) | 1/49 | 1/36
Fever > 39°C but ≤ 40°C (General disorders) | 0/49 | 0/36
Fever > 40°C (General disorders) | 0/49 | 0/36
Decreased appetite (General disorders) | 6/49 | 4
Irritability (General disorders) | 9/49 | 4/35
Increased sleep (General disorders) | 2 | 5
Decreased sleep (General disorders) | 0/48 | 2
Rash (General disorders) | 3 | 1

LIMITATIONS AND CAVEATS:
Primary analysis based on evaluable immunogenicity population as per analysis plan change.Data for a participant reported in PCV/23vPS/13vPnC instead of PCV/PCV/13vPnC due to data entry error on case report form;this did not affect result conclusion.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.